CLINICAL TRIAL: NCT02757092
Title: The Efficacy of Home-Based Pulmonary Rehabilitation Training in Aged Patients With Lung Tumor After Video-assisted Thoracic Surgery:A Clinical Randomized Trial
Brief Title: The Impacts of Pulmonary Rehabilitation Therapy on Patients After Thoracic Surgery
Acronym: VATSMIPMEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Liu Jui Fang, Respiratory therapist, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1046659A3
Record Dates: First submitted 2016-04-12; First posted 2016-04-29 (Estimated); Results first posted 2020-11-03 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Lung Neoplasms
Keywords: Pulmonary rehabilitation; surgery; exercise
MeSH Terms: conditions — Lung Neoplasms; Motor Activity

STUDY DESIGN:
Intervention Model Description: This study employed a prospective, randomized, and controlled clinical design to determine the efficacy of home-based pulmonary rehabilitation in patients after thoracoscopy. After participants signed the consent form, they were randomly included into the control or experimental group on the day of discharge. The random assignment was performed based on simple randomization by using numbers from 1 to 36; numbered, sealed, opaque envelopes were used for allocation concealment. These envelopes were randomly distributed by non researchers and recorded.
Who Masked: Participant
Masking Description: After participants signed the consent form, they were randomly included into the control or experimental group on the day of discharge
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Home-based rehabilitation program (Experimental): 0-2 weeks,1. aerobic exercise intensity was targeted to reach 10-11 points of perceived exercise (RPE) scale 2. raised their upper limbs while simultaneously performing lower-limb stepping at place for 20 min 3.walked at a comfortable speed for 15 min twice per day.4. Triflo-II was performed 8-10 times per hour. inspiratory muscle training with the initial pressure set at 25%-30% of the maximum inspiratory pressure.3-6 weeks, aerobic exercise reach 12-15 points on the RPE scale. upper-limb resistance exercise (raising of a 250-cc water bottle) and lower-limb stepping for 20 min per day , walking exercise for a total of 30 min. Triflo-II was performed 8-10 times per hour, and train the inspiratory muscle with the pressure intensity adjusted to more than 5% of that in the first stage.
  Interventions: Other: Home-based Pulmonary Rehabilitation
- standard care (Active Comparator): control group accept the pulmonary rehabilitation (breathing exercise, extremities exercise, breathing muscle training, incentive spirometry (Triflo-II) training, intermittent positive pressure ventilation, chest physical therapy and pain control) only in operation stage on before op-day 3 day and after op-day and without home based pulmonary rehabilitation.
  Interventions: Other: Home-based Pulmonary Rehabilitation

INTERVENTIONS:
Other: Home-based Pulmonary Rehabilitation — (1) breathing exercises (pursed-lip and diaphragmatic breathing) and coughing exercises, (2) aerobic exercises (upper and lower limb exercises and walking), (3) incentive spirometry training (Triflo-II), and (4) threshold load training of the inspiratory muscle. In the first stage (0-2 weeks), the aerobic exercise intensity was targeted to reach 10-11 points on the 20-point Borg rating of perceived exercise (RPE) scale. Patients raised their upper limbs while simultaneously performing lower-limb stepping at place for 20 min; in addition, they walked at a comfortable speed for 15 min twice per day. Incentive spirometry training (Triflo-II) was performed 8-10 times per hour. We used a threshold load trainer for inspiratory muscle training (30 breaths each time, twice per day) with the initial pressure set at 25%-30% of the maximum inspiratory pressure.

SUMMARY:
The advantages of thoracoscopic surgery include smaller wounds, fewer postoperative complications, and shortened hospital stay. However,complications such as pain, pulmonary function insufficiency, pneumonia,postoperative pneumothorax, persistent air leakage, subcutaneous emphysema, cough, and hemoptysis may occur in older patients after thoracoscopic surgery. Pulmonary rehabilitation has been demonstrated by evidence-base medicine could effectively reduce pulmonary complications and dyspnea as well as improve lung function, quality of life, exercise ability, and functional status of patients after traditional heart and thoracic surgery. Studies have suggested that pulmonary rehabilitation should be performed for at least 4 weeks to optimize the training effect .However, most patients who undergo thoracoscopic surgery were discharged within 3-5 days. Such a short hospital stay impeded the delivery of pulmonary rehabilitation. Home-based pulmonary rehabilitation appeared to be an option for these patients The purpose of this study is to determine whether Pulmonary rehabilitation are effective on patients who had thoracic surgeries.

DETAILED DESCRIPTION:
Pulmonary-related surgeries remain some potential risks according to the previous evidence-based studies. Particularly, individuals who were over 65 years of age with smoking, chronic pulmonary disease, wheezy, cardiovascular comorbidities, upper respiratory infection were at the high risk of pulmonary complications after surgery,which accounted for approximately 2% to 40% of occurrence rate. The average mortality rate due to surgery was approximately 2%-8% in patients aged more than 65 years.Pulmonary rehabilitation could effectively reduce pulmonary complications and dyspnea as well as improve lung function, quality of life, exercise ability, and functional status of patients after traditional heart and thoracic surgery.But efficacy of home-based pulmonary rehabilitation for older adults following thoracoscopic surgery, it has not received much attention.

This study employed a prospective, randomized, and controlled clinical design to determine the efficacy of home-based pulmonary rehabilitation in older adults after VATS. All participants underwent preoperative and initial postoperative pulmonary rehabilitation during their hospital stay and were randomly assigned to the experimental or control group at the time of discharge. The control group received standard health education, whereas the experimental group received home-based pulmonary rehabilitation in addition to standard health education. Objective and personal subjective outcome measurements were performed before hospital discharge and 2, 6, and 12 weeks after discharge The control group received standard care. Considering the principle for exercise progression, we divided the home-based rehabilitation program into two stages (0-2 weeks and 3-6 weeks).The exercise program was adjusted in the second week when patients visited the outpatient department of the hospital for follow-up. The home-based rehabilitation program included (1) breathing exercises (pursed-lip and diaphragmatic breathing) and coughing exercises, (2) aerobic exercises (upper and lower limb exercises and walking), (3) incentive spirometry training (Triflo-II), and (4) threshold load training of the inspiratory muscle. In the first stage (0-2 weeks), the aerobic exercise intensity was targeted to reach 10-11 points on the 20-point Borg rating of perceived exercise (RPE) scale. Patients raised their upper limbs while simultaneously performing lower-limb stepping at place for 20 min; in addition, they walked at a comfortable speed for 15 min twice per day. Incentive spirometry training (Triflo-II) was performed 8-10 times per hour. We used a threshold load trainer for inspiratory muscle training (30 breaths each time, twice per day) with the initial pressure set at 25%-30% of the maximum inspiratory pressure.

In the second stage (3-6 weeks), the aerobic exercise intensity was targeted to reach 12-15 points on the RPE scale. Patients performed upper-limb resistance exercise (raising of a 250-cc water bottle) and lower-limb stepping for 20 min per day as well as walking exercise (slow walking for 5 min and fast walking for 2 min, followed by 5-min slow walking, for a total of 30 min). Incentive spirometry training (Triflo-II) was performed 8-10 times per hour, and a threshold load trainer was used to train the inspiratory muscle (30 breaths each time, twice per day), with the pressure intensity adjusted to more than 5% of that in the first stage.Researchers contacted patients at home every week through phone calls to monitor the occurrence of any uncomfortable reaction and to encourage patients to continue their rehabilitation program.

ELIGIBILITY:
Inclusion Criteria:

1. Signed consent
2. The men and women over the age of 65
3. admission to undergo VATS.
4. consciousness and ability to communicate
5. ability to undergo 6 weeks of a home-based pulmonary rehabilitation program

Exclusion Criteria:

1. refusal to participate
2. unplanned emergency surgery
3. hemodynamic instability
4. received other surgery within a month postsurgery
5. unconsciousness after surgery
6. bedridden and upper or lower limb weakness
7. received radiation and chemotherapy postsurgery
8. implementation of thoracoscopic surgery for biopsy only

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-03-31 (Actual); Primary Completion 2017-04-01 (Actual); Study Completion 2017-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jui Fang Liu, PhD, Study Director — Department of Respiratory Therapy; Nai Ying Kuo, master, Study Chair — Department of Respiratory Therapy
Locations (2):
- Taiwan (2):
  - Chang Gung Memorial Hospital, Kaohsiung City, Niaosong
  - Chang Gung Memorial Hospital, Kaohsiung City

IPD SHARING:
Plan to Share IPD: Yes
Share Protocol and Outcome deta
Supporting Information: Study Protocol, CSR
Time Frame: starting 6 months after publication
Access Criteria: connect with miss Nai ying kuo and Share IPD by email

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was design a Prospective randomized control trial,and enrolled a total of 36 older patients with lung tumors after thoracoscopic surgery in the cardiothoracic and vascular ordinary ward between March 31 2016 to April 1 2017. The study was performed conducted in Kaohsiung Chang Gung Memorial Hospital, Taiwan
Groups:
- Home Pulmonary Rehabilitation Group: Pulmonary Rehabilitation group accept the pulmonary rehabilitation( breathing exercise, extremities exercise, breathing muscle training, incentive spirometry (Triflo-II) training, intermittent positive pressure ventilation, chest physical therapy ) in operation stage on before op-day 3 day and after op-day 2 weeks and keep home based pulmonary rehabilitation on discharge 2 weeks, 6 weeks and after 12 weeks.
  study group : received pain medication and standard care
- Study Group: study group accept the pulmonary rehabilitation( breathing exercise, extremities exercise, breathing muscle training, incentive spirometry (Triflo-II) training, intermittent positive pressure ventilation, chest physical therapy ) in operation stage on before op-day 3 day and after op-day ,after discharged received standard care
Period: Overall Study
Arm/Group | Home Pulmonary Rehabilitation Group | Study Group
Started | 18 (Random assignment was to encode subjects from opaque envelopes and sealed, on the day of discharge) | 18 (Random assignment was to encode subjects from opaque envelopes and sealed, on the day of discharge)
Completed | 18 (All subjects completed the study) | 18 (All subjects completed the study)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Pearson chi-square test was used for sex. comorbidities and smoking, Student's t-test was used for age, body weight . Body Mass Index, and total hospital days, Data is presented as either n(%) or mean ± SD.
Groups:
- Pulmonary Rehabilitation Group: arm group accept the pulmonary rehabilitation( smoking cession before operation, breathing exercise, extremities exercise, breathing muscle training, incentive spirometry (Triflo-II) training, intermittent positive pressure ventilation, chest physical therapy and pain control) in operation stage on before op-day 3 day and after op-day 2 weeks and keep home based pulmonary rehabilitation on discharge 2 weeks, 6 weeks and after 12 weeks.
- The Control Group: The control group received pain medication and usual care.
- Total: Total of all reporting groups
Arm/Group | Pulmonary Rehabilitation Group | The Control Group | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Categorical [Count of Participants; unit: Participants] — After signing the consent form, each case subject was randomly divided assigned into either the control or the experimental group on the day of discharge.Inclusion criteria were: 1) Older than or equal to 65 years with an established diagnosis of Lung tumor.2)admission to receive video-assisted thoracoscopic surgery 3.)conscious and able to communicate, and 4.)Able to undergo six weeks of home-based pulmonary rehabilitation program.
  Participants
    Count of Participants: <=18 years | 0 | 0 | 0
    Count of Participants: Between 18 and 65 years | 0 | 0 | 0
    Count of Participants: >=65 years | 18 | 18 | 36
Sex: Female, Male [Count of Participants; unit: Participants] — Pearson chi-square test was used for sex,deta is presented as either n(%) or mean +-SD
  Participants
    Female | 8 | 11 | 19
    Male | 10 | 7 | 17
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants] — enrolled a total of 36 older patients with lung tumors after thoracoscopic surgery in the cardiothoracic and vascular ordinary ward in Taiwan
  Participants
    Taiwan | 18 | 18 | 36
BMI (Kg/m2) [Mean (Standard Deviation); unit: Kg/m2] — Student's t-test was used for Body Mass Index .Data is presented as either n(%) or mean ± SD.
  Kg/m2 | 25.08 (3.3) | 23.46 (2.8) | 24.27 (3.05)
BW (kg) [Mean (Standard Deviation); unit: kg] — Student's t-test was used for body weight. Data is presented as either n(%) or mean ± SD.
  kg | 65.33 (11.71) | 57.98 (9.44) | 61.66 (10.57)
Amount of comorbidities [Count of Participants; unit: Participants] — Pearson chi-square test was used for sex. comorbidities and smoking, Data is presented as either n(%) or mean ± SD.
  Participants
    Hypertension | 7 | 11 | 18
    DM | 5 | 4 | 9
    Cardiovascular diseases n | 2 | 4 | 6
    COPD | 9 | 2 | 11
smoking [Count of Participants; unit: Participants] | 6 | 4 | 10
total hospital days [Mean (Standard Deviation); unit: days] — Student's t-test was used for total hospital days, Data is presented as either n(%) or mean ± SD
  days | 8.68 (4.41) | 8.32 (3.28) | 8.5 (3.85)
PFT [Mean (Standard Deviation); unit: liter/sec] — Student's t-test was used for FVC .Data is presented as either n(%) or mean ± SD.
  liter/sec
    FEV1(liter/sec) | 1.88 (0.44) | 1.78 (0.93) | 1.83 (0.69)
    FVC(liter/sec) | 1.48 (0.47) | 1.43 (0.71) | 1.45 (0.59)
    MMEF25-75(liter/sec) | 1.80 (1.17) | 1.41 (0.77) | 1.61 (0.97)
    PEFR(liter/sec) | 4.08 (2.05) | 3.01 (1.46) | 3.55 (1.76)
FEV1/FVC(%) [Mean (Standard Deviation); unit: %] — Measure Description: Student's t-test was used for FEV1/FVC(%).Data is presented as either n(%) or mean ± SD.The FEV1/FVC ratio is a calculated ratio used in the diagnosis of obstructive and restrictive lung disease. It represents the proportion of a person's vital capacity that they are able to expire in the first second of forced expiration (FEV1) to the full, forced vital capacity (FVC) The result of this ratio is expressed as FEV1%.Normal values are approximately 75%.values less than 0.70 are suggestive of airflow limitation with an obstructive pattern
  % | 79.02 (17.01) | 81.03 (10.45) | 80.03 (13.73)
Modified Borg score [Mean (Standard Deviation); unit: scores on a scale] — Student's t-test was used for Modified Borg score .Data is presented as mean ± SD.Scores on a scale that ranges from 1 to 10,Larger numbers indicate more severe breathing difficulties,the opposite is the smaller the number, the lower the dyspnea is
  scores on a scale | 1.61 (0.6) | 1.89 (0.58) | 1.75 (0.59)
MIP(cmH2O) [Mean (Standard Deviation); unit: cmH2O] — Student's t-test was used for MIP/MEP Data is presented as either n(%) or mean ± SD.
  cmH2O | 50.22 (11.89) | 49.73 (16.83) | 49.98 (13.82)
MEP(cmH2O) [Mean (Standard Deviation); unit: cmH20] — Student's t-test was used for MIP/MEP Data is presented as either n(%) or mean ± SD.
  cmH20 | 61.89 (24.00) | 50.40 (21.06) | 56.15 (23.36)
Lung capacity (mL/sec) [Mean (Standard Deviation); unit: mL] — Lung capacity measure by incentive spirometry (Triflow) , The flow-oriented incentive spirometer (Triflow device) consists of three chambers in series, each of which contains a ball.An inspiratory flow of 600 mL/sec is required to raise the first ball, an inspiratory flow of 900 mL/sec is required to elevate the first and second balls, and a flow of 1200 mL/sec is required to elevate all three balls.The time of the ball stays longer was mean the better lung capacity
  mL | 1200.00 (534.68) | 1000.00 (524.68) | 1100.00 (529.68)
6-min walk test(meter,M) [Mean (Standard Deviation); unit: meter] — The 6MWT is a useful measure of functional capacity targeted at people with at least moderately severe impairment. The test has been widely used for preoperative and postoperative evaluation and for measuring the response to therapeutic interventions for pulmonary and cardiac disease.In healthy subjects, the 6-min walk distance (6MWD) ranges from 400 to 700 m, the main predictor variables being gender, age and height.The longer distance was mean the better functional capacity ability,<250 m does predict poorer outcome
  meter | 364.33 (49.89) | 315.22 (59.34) | 339.78 (54.62)
Anesthesia time(min) [Mean (Standard Deviation); unit: min] — Student's t-test was used for Anesthesia time
  min | 271.15 (83.52) | 249.84 (70.83) | 260.5 (77.18)
American Society of Anesthesiologists (ASA) score [Mean (Standard Deviation); unit: scores on a scale] — Student's t-test was used for ASA score. Data is presented as mean ± SD.Scores on a scale that ranges from 1 to 6. ASA 1: A normal healthy patient. ASA 2: A patient with a mild systemic disease. ASA 3: A patient with a severe systemic disease that is not life-threatening. ASA 4: A patient with a severe systemic disease that is a constant threat to life. ASA 5: A moribund patient who is not expected to survive without the operation. ASA 6: A brain-dead patient whose organs are being removed with the intention of transplanting them into another patient.
  scores on a scale | 2.11 (0.32) | 2.11 (0.58) | 2.11 (0.45)
Surgery time(min) [Mean (Standard Deviation); unit: min] — Student's t-test was used for Surgery time , Data is presented as either n(%) or mean ± SD.
  min | 236.90 (79.02) | 225.26 (66.32) | 231.08 (72.67)
chest tube placement time(hours) [Mean (Standard Deviation); unit: hours] — Student's t-test was used for Chest tube placement time, Data is presented as either n(%) or mean ± SD.
  hours | 115.05 (37.56) | 118.11 (50.90) | 116.58 (44.23)
surgery method [Count of Participants; unit: Participants]
  lobectomy | 11 | 12 | 23
  wedge resection | 5 | 5 | 10
  sefmentectomy | 2 | 1 | 3
wedge resection [Count of Participants; unit: Participants] | 5 | 5 | 10
surgery site [Count of Participants; unit: Participants] — Pearson chi-square test was used for surgery site. Data is presented as either n(%) or mean ± SD. Some patients have operation two lobes at the same time, so the total is not necessarily equal to 18.
  Participants
    Right upper lobe | 12 | 7 | 19
    Right middle lobe | 1 | 1 | 2
    Right low lobe | 3 | 4 | 7
    left upper lobe | 0 | 5 | 5
    left low lobe | 3 | 1 | 4
postoperative diagnosis [Count of Participants; unit: Participants] — Pearson chi-square test was used for postoperative diagnosis.Data is presented as either n(%) or mean ± SD.
  Participants
    small cell carcinoma | 1 | 0 | 1
    adenocarcinoma | 14 | 13 | 27
    large cell carcinoma | 1 | 0 | 1
    sguamous cell carcinoma | 0 | 3 | 3
    benign lung tumor | 2 | 2 | 4
postoperative stages of lung cancer [Count of Participants; unit: Participants] — Pearson chi-square test was used postoperative stages of lung cancer. Surgery time and Chest tube placement time, Data is presented as either n(%) or mean ± SD.StageI:Cancer may be present in the underlying lung tissues, but the lymph nodes remain unaffected. StageII:The cancer may have spread to nearby lymph nodes or into the chest wall.StageIII:The cancer is continuing to spread from the lungs to the lymph nodes or to nearby structures and organs.Stage IV: the cancer has metastasized, or spread, beyond the lungs into other areas of the body,the last stages of cancer means the more serious
  Participants
    stage1 n(%) | 11 | 8 | 19
    stage2 n(%) | 4 | 7 | 11
    Benign lung tumor(%) | 2 | 2 | 4
    others,ground-glass opacity(%) | 1 | 1 | 2
postoperative complications [Count of Participants; unit: Participants]
  emphysema | 16 | 15 | 31
  air leak | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Discharge 2weeks Exercise Capacity
Description: Exercise capacity as assessed by 6 min walking test(M).The 6-min walk test (6 MWT) is a submaximal exercise test that entails measurement of distance walked over a span of 6 minutes. The 6-minute walk distance (6 MWD) provides a measure for integrated global response of multiple cardiopulmonary and musculoskeletal systems involved in exercise . The 6 MWT provides information regarding functional capacity, response to therapy and prognosis across a broad range of chronic cardiopulmonary conditions .The normal range in aged patients 60-69 y(male 572 m,female 538 M),70-79 y(male 527 m,female 471 M),80-89 y(male 417 m,female 392 M)higher scores mean a better outcome.
Time Frame: assessed at discharge 2weeks
Population: 2-WAY repeated measures ANOVA method was used for exercise capacity.an intention-to-treat analysis was performed.group × time interactions were observed for the 6-min walking distance.
Measure: Mean (Standard Deviation); unit: meter(M)
Groups:
- Pulmonary Rehabilitation Group 2 Weeks Six-min Walking Distanc; The Control Group 2weeks Six-min Walking Distanc: Each subject received six-min walking distance assessments at discharge 2 weeks after discharge
Arm/Group | Pulmonary Rehabilitation Group 2 Weeks Six-min Walking Distanc | The Control Group 2weeks Six-min Walking Distanc
Number analyzed (Participants) | 18 | 18
meter(M) | 408.61 (62.85) | 311.94 (84.65)
Statistical Analysis 1: Comparison: Pulmonary Rehabilitation Group 2 Weeks Six-min Walking Distanc vs The Control Group 2weeks Six-min Walking Distanc; Test type: Superiority; p < 0.05, ANOVA

2. Primary Outcome: Discharge 6 Weeks Exercise Capacity
Description: as for outcome 1
Time Frame: assessed at discharge.6weeks
Population: 2-WAY repeated measures ANOVA method was used for exercise capacity. For group comparisons, an intention-to-treat analysis was performed.group × time interactions were observed for the 6-min walking distance.
Measure: Mean (Standard Deviation); unit: meter(M)
Groups:
- Pulmonary Rehabilitation Group 6 Weeks Six-min Walking Distanc: Each subject received six-min walking distance assessments at 6 weeks after discharge
- The Control Group 6 Weeks Six-min Walking Distanc: Each subject received six-min walking distance assessments at discharge6 weeks, after discharge
Arm/Group | Pulmonary Rehabilitation Group 6 Weeks Six-min Walking Distanc | The Control Group 6 Weeks Six-min Walking Distanc
Number analyzed (Participants) | 18 | 18
meter(M) | 411.63 (44.49) | 332.94 (54.03)
Statistical Analysis 1: Comparison: Pulmonary Rehabilitation Group 6 Weeks Six-min Walking Distanc vs The Control Group 6 Weeks Six-min Walking Distanc; null hypothesis; Test type: Superiority; p < 0.05, ANOVA

3. Primary Outcome: Discharge 12 Weeks Exercise Capacity
Description: Exercise capacity as assessed by 6 min walking test(M).The 6-min walk test (6 MWT) is a submaximal exercise test that entails measurement of distance walked over a span of 6 minutes. The 6-minute walk distance (6 MWD) provides a measure for integrated global response of multiple cardiopulmonary and musculoskeletal systems involved in exercise . The 6 MWT provides information regarding functional capacity, response to therapy and prognosis across a broad range of chronic cardiopulmonary conditions .The normal range in aged patients 60-69 y(male 572 m,female 538 M),70-79 y(male 527 m,female 471 M),80-89 y(male 417 m,female 392 M).higher scores mean a better outcome.
Time Frame: assessed at discharge 12 weeks
Population: 2-WAY repeated measures ANOVA method was used for exercise capacity. For group comparisons, an intention-to-treat analysis was performed. group × time interactions were observed for the 6-min walking distance.
Measure: Mean (Standard Deviation); unit: meter(M)
Groups:
- Pulmonary Rehabilitation group12 Weeks Six-min Walking Distanc; The Control Group 12 Weeks Six-min Walking Distanc: Each subject received six-min walking distance assessments at discharge 12 weeks after discharge
Arm/Group | Pulmonary Rehabilitation group12 Weeks Six-min Walking Distanc | The Control Group 12 Weeks Six-min Walking Distanc
Number analyzed (Participants) | 18 | 18
meter(M) | 397.06 (50.37) | 345.17 (46.04)
Statistical Analysis 1: Comparison: Pulmonary Rehabilitation group12 Weeks Six-min Walking Distanc vs The Control Group 12 Weeks Six-min Walking Distanc; Test type: Superiority; p < 0.05, ANOVA

4. Secondary Outcome: Discharge 2 Weeks Forced Vital Capacity (FVC in Liter(L)/Sec)
Description: Forced vital capacity (FVC in L/sec) assessment by pulmonary function test.Normal values in healthy males aged 20-60 from 4.5-3.5 L/sec,and for females from 3.25-2.5 L/sec ,and whether higher scores mean a better outcome.
Time Frame: assessments at 2 weeks after discharge
Population: 2-WAY repeated measures ANOVA method was used for pulmonary function test.
Measure: Mean (Standard Deviation); unit: liter(L)/sec
Groups:
- Pulmonary Rehabilitation Group 2 Weeks FVC (Liter(L)/Sec): Each subject received FVC assessments at 2 weeks after discharge
- The Control Group 2 Weeks FVC(Liter(L)/Sec)): Each subject received FVC assessments at 2 weeks discharge
Arm/Group | Pulmonary Rehabilitation Group 2 Weeks FVC (Liter(L)/Sec) | The Control Group 2 Weeks FVC(Liter(L)/Sec))
Number analyzed (Participants) | 18 | 18
liter(L)/sec | 2.48 (0.80) | 2.00 (0.85)
Statistical Analysis 1: Comparison: Pulmonary Rehabilitation Group 2 Weeks FVC (Liter(L)/Sec) vs The Control Group 2 Weeks FVC(Liter(L)/Sec)); Test type: Superiority; p < 0.05, ANOVA

5. Secondary Outcome: Discharge 2weeks Forced Expiratory Volume in 1 Second(FEV1,Liter(L)/Sec)
Description: The Forced Expiratory Volume in 1 Second parameter measures the volume of air that was exhaled into the mouthpiece in the first second after a full inhalation. The Measured column represents the total volume exhaled during the first second, in liters. Normal values in healthy males aged 20-60 range from 4.5 to 3.5 liters, and normal values for females aged 20-60 range from 3.25 to 2.5 liters. The Predicted column compares the actual volume breathed out during the first second of your test to an average of the normal volume breathed out in 1 second for a person of the same gender, height, and age. This value is expressed as a percentage, with normal test values being between 80% and 120% of the average (predicted) values.and whether higher scores mean a better outcome.
Time Frame: assessed at 2 weeks after discharge
Population: 2-WAY repeated measures ANOVA method was used for pulmonary function test.
Measure: Mean (Standard Deviation); unit: liter(L)/sec
Groups:
- Pulmonary Rehabilitation Group 2 Weeks FEV1 (Liter(L)/Sec): Each subject received FEV1 (liter(L)/sec)assessments at 2 weeks after discharge
- The Control Group 2 Weeks FEV1(Liter(L)/Sec): Each subject received FEV1(liter(L)/sec) assessments at 2 weeks after discharge
Arm/Group | Pulmonary Rehabilitation Group 2 Weeks FEV1 (Liter(L)/Sec) | The Control Group 2 Weeks FEV1(Liter(L)/Sec)
Number analyzed (Participants) | 18 | 18
liter(L)/sec | 1.97 (0.54) | 1.57 (0.69)
Statistical Analysis 1: Comparison: Pulmonary Rehabilitation Group 2 Weeks FEV1 (Liter(L)/Sec) vs The Control Group 2 Weeks FEV1(Liter(L)/Sec); Test type: Superiority; p < 0.05, ANOVA

6. Secondary Outcome: Discharge 2weeks MMEF 25-75%(Liter(L)/Sec)
Description: Forced expiratory flow (FEF) is the flow (or speed) of air coming out of the lung during the middle portion of a forced expiration. It can be given at discrete times, generally defined by what fraction of the forced vital capacity (FVC) has been exhaled. The usual discrete intervals are 25%, 50% and 75%, usually 25-75% (FEF25-75%).Predicted normal values for FEF depend on age, sex, height, mass and ethnicity as well as the research study that they are based on assessment by pulmonary function test and higher scores mean a better outcome.
Time Frame: assessed at discharge 2weeks
Population: 2-WAY repeated measures ANOVA method was used for pulmonary function test.
Measure: Mean (Standard Deviation); unit: liter(L)/sec
Groups:
- Pulmonary Rehabilitation Group; The Control Group: Each subject received MMEF25-75%(liter(L)/sec) assessments at 2 weeks after discharge
Arm/Group | Pulmonary Rehabilitation Group | The Control Group
Number analyzed (Participants) | 18 | 18
liter(L)/sec | 2.00 (0.81) | 1.58 (0.94)
Statistical Analysis 1: Comparison: Pulmonary Rehabilitation Group vs The Control Group; null hypothesis; Test type: Superiority; p < 0.05, ANOVA

7. Secondary Outcome: Discharge 2weeks Peak Expiratory Flow Rate(PEFR , Liter(L)/Sec)
Description: Peak expiratory flow rate (PEFR in liter(L)/sec) assessment by pulmonary function test.It measures the airflow through the bronchi and thus the degree of obstruction in the airways. Peak expiratory flow is typically measured in units of liters per second (L/sec).when measured as part of spirometry.The normal range 500-700 L/sec In men, for women, the normal range is 380-500 L/sec.higher scores mean a better outcome.
Time Frame: assessed at discharge 2weeks
Population: 2-WAY repeated measures ANOVA method was used for pulmonary function test.
Measure: Mean (Standard Deviation); unit: liter(L)/sec
Groups:
- Pulmonary Rehabilitation Group; The Control Group: Each subject received PEFR assessments at 2 weeks after discharge
Arm/Group | Pulmonary Rehabilitation Group | The Control Group
Number analyzed (Participants) | 18 | 18
liter(L)/sec | 5.68 (2.35) | 4.27 (2.35)
Statistical Analysis 1: Comparison: Pulmonary Rehabilitation Group vs The Control Group; null hypothesis; Test type: Superiority; p < 0.05, ANOVA

8. Secondary Outcome: Discharge 2weeks Inspiratory Muscle Strength(MIP,cmH2O)
Description: Inspiratory muscle strength as assessed by Maximum inspiratory pressure (MIP, cmH2O).The MIP is a measure of inspiratory muscle strength produced by a sub-atmospheric pressure The normal.range of MIP in elderly people approximately 60 cm H2O for men and 40 cm H2O for women .An absolute MIP value of < - 40 cm H2O is always abnormal,and higher scores was mean a better outcome.
Time Frame: assessed at discharge 2 weeks.
Population: Two-way repeated measures ANOVA for MIP. For group comparisons, an intention-to-treat analysis was performed. group × time interactions were observed for the MIP
Measure: Mean (Standard Deviation); unit: cmH2O
Groups:
- Pulmonary Rehabilitation Group 2 Weeks MIP(cmH2O); The Control Group 2weeks MIP (cmH2O): Each subject received MIP assessments at discharge, and 2 weeks, 6 weeks, and 12 weeks after discharge
Arm/Group | Pulmonary Rehabilitation Group 2 Weeks MIP(cmH2O) | The Control Group 2weeks MIP (cmH2O)
Number analyzed (Participants) | 18 | 18
cmH2O | 90.00 (25.66) | 67.33 (28.15)
Statistical Analysis 1: Comparison: Pulmonary Rehabilitation Group 2 Weeks MIP(cmH2O) vs The Control Group 2weeks MIP (cmH2O); Test type: Superiority; p < 0.05, ANOVA

9. Secondary Outcome: Discharge 2weeks Expiratory Muscle Strength(MEP,cmH2O)
Description: The Maximal Expiratory Pressure (MEP) are global measures of the maximal strength of the respiratory muscles.(MEP, cmH2O) .MEP is a supra-atmospheric pressure which can be developed in an effort of the abdominal and intercostal muscles.Expiratory muscle strength assesses extrathoracic muscle health.An absolute MEP value of < 80 cmH2O is always abnormal, and higher scores mean a better outcome.
Time Frame: assessed at discharge 2 weeks
Population: Two-way repeated measures ANOVA for MEP. an intention-to-treat analysis was performed.group × time interactions were observed for the MEP
Measure: Mean (Standard Deviation); unit: cmH2O
Groups:
- Pulmonary Rehabilitation Group 2 Weeks MEP(cmH2O); The Control Group 2weeks MEP(cmH2O): Each subject received MEP assessments at discharge, and 2 weeks, 6 weeks, and 12 weeks after discharge
Arm/Group | Pulmonary Rehabilitation Group 2 Weeks MEP(cmH2O) | The Control Group 2weeks MEP(cmH2O)
Number analyzed (Participants) | 18 | 18
cmH2O | 89.44 (28.79) | 68.89 (22.72)
Statistical Analysis 1: Comparison: Pulmonary Rehabilitation Group 2 Weeks MEP(cmH2O) vs The Control Group 2weeks MEP(cmH2O); Test type: Superiority; p < 0.05, ANOVA

10. Secondary Outcome: Discharge 2 Weeks Modified Borg Score
Description: Dyspnea score as assessed by Modified Borg score, The literature review clearly showed that the Modified Borg score was a valid and reliable tool when used in pulmonary medicine and in exercise physiology studies.The scale used was perceived exertion adapted to be appropriate for measuring dyspnea. This consisted of a vertical scale labelled 0-10, with corresponding verbal expressions of progressively increasing perceived sensation intensity. It starts at number 0 that mean breathing is no difficulty at all and progresses through to number 10 that mean breathing difficulty is maximal.so higher scores mean a worse outcome
Time Frame: assessed at discharge 2 weeks
Population: Two-way repeated measures ANOVA for Modified Borg score.an intention-to-treat analysis was performed.group × time interactions were observed for the Modified Borg score
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- Pulmonary Rehabilitation Group 2 weeksModified Borg Score; The Control Group 2weeks Modified Borg Score: Each subject received Modified Borg score assessments at discharge, and 2 weeks, 6 weeks, and 12 weeks after discharge
Arm/Group | Pulmonary Rehabilitation Group 2 weeksModified Borg Score | The Control Group 2weeks Modified Borg Score
Number analyzed (Participants) | 18 | 18
scores on a scale | 1.06 (0.54) | 1.72 (0.67)
Statistical Analysis 1: Comparison: Pulmonary Rehabilitation Group 2 weeksModified Borg Score vs The Control Group 2weeks Modified Borg Score; Test type: Superiority; p < 0.05, ANOVA

11. Secondary Outcome: Discharge 2weeks Lung Expansion Capacity
Description: Lung expansion capacity as assessed by incentive spirometry with the flow-oriented device( Triflow II,volume × seconds) (ml).Incentive spirometry that feedback respiratory training can improve respiratory function, endurance for exercise capacity,Wide flow rate range from 600 - 1200(volume × seconds) (ml).higher scores mean a better outcome.
Time Frame: assessed at discharge 2 weeks
Population: Two-way repeated measures ANOVA for Lung expansion capacity. an intention-to-treat analysis was performed.group × time interactions were observed for the Lung expansion capacity.
Measure: Mean (Standard Deviation); unit: (ml)
Groups:
- Pulmonary Rehabilitation: study group follow Triflo on discharge 2 weeks
- Control Group: control group follow Triflo on discharge 2 weeks
Arm/Group | Pulmonary Rehabilitation | Control Group
Number analyzed (Participants) | 18 | 18
(ml) | 1450.00 (619.53) | 1033.33 (388.65)
Statistical Analysis 1: Comparison: Pulmonary Rehabilitation vs Control Group; Test type: Superiority; p < 0.05, ANOVA

12. Secondary Outcome: Postoperative 2 Weeks Pulmonary Complications
Description: Pulmonary complication as assessed by Chest X-ray.pneumonia.lung collapse.atelectasis.emphysema and pleural effusion were collected.some patients have two pulmonary complications at the same time, such as emphysem and infiltration, so the total number is not necessarily equal to 18.
Time Frame: at 2weeks after discharge
Population: Pearson chi-square test was used for Pulmonary complication on discharge 2 weeks .Data is presented as either n(%).
Measure: Count of Participants; unit: Participants
Groups:
- Pulmonary Rehabilitation: study group follow CXR on discharge 2 weeks
- Control Group: control group follow CXR on discharge 2 weeks
Arm/Group | Pulmonary Rehabilitation | Control Group
Number analyzed (Participants) | 18 | 18
Participants
  pneumonia | 0 | 1
  atelectasis | 1 | 2
  pleural effusion | 0 | 1
  emphysema | 0 | 1
  pulmonary infilation | 1 | 0
Statistical Analysis 1: Comparison: Pulmonary Rehabilitation vs Control Group; Descriptive statistics were expressed as mean ± standard deviation or median and interquartile range depending on the nature and distribution of the variables; Test type: Superiority; p = 0.05, Chi-squared

13. Secondary Outcome: Discharge 6 Weeks Forced Vital Capacity(Liter(L)/Sec)
Description: Forced vital capacity (FVC in (liter(L)/sec)) assessment by pulmonary function test.Normal values in healthy males aged 20-60 from 4.5-3.5 (liter(L)/sec),and for females from 3.25-2.5 (liter(L)/sec) ,and whether higher scores mean a better outcome.
Time Frame: assessments at discharge 6 weeks
Population: 2-WAY repeated measures ANOVA method was used for pulmonary function test.
Measure: Mean (Standard Deviation); unit: liter( L)/sec
Groups:
- Pulmonary Rehabilitation Group 6 Weeks FVC(Liter(L)/Sec): Each subject received (FVC in liter(L)/sec) assessments at 6 weeks after discharge
- The Control Group 6 Weeks FVC (Liter(L)/Sec): Each subject received FVC assessments at 6 weeks after discharge
Arm/Group | Pulmonary Rehabilitation Group 6 Weeks FVC(Liter(L)/Sec) | The Control Group 6 Weeks FVC (Liter(L)/Sec)
Number analyzed (Participants) | 18 | 18
liter( L)/sec | 2.48 (0.88) | 1.97 (0.80)
Statistical Analysis 1: Comparison: Pulmonary Rehabilitation Group 6 Weeks FVC(Liter(L)/Sec) vs The Control Group 6 Weeks FVC (Liter(L)/Sec); null hypothesis; Test type: Superiority; p < 0.05, ANOVA

14. Secondary Outcome: Discharge 6 Weeks Forced Expiratory Volume in 1 Second (FEV1,Liter(L)/Sec)
Description: as for outcome 5
Time Frame: assessed at discharge 6weeks
Population: 2-WAY repeated measures ANOVA method was used for pulmonary function test.
Measure: Mean (Standard Deviation); unit: liter(L)/sec
Groups:
- Pulmonary Rehabilitation Group 6 Weeks FEV1,Liter(L)/Sec; The Control Group 6 Weeks FEV1,Liter(L)/Sec: Each subject received FEV1 assessments at discharge 6 weeks after discharge
Arm/Group | Pulmonary Rehabilitation Group 6 Weeks FEV1,Liter(L)/Sec | The Control Group 6 Weeks FEV1,Liter(L)/Sec
Number analyzed (Participants) | 18 | 18
liter(L)/sec | 2.02 (0.60) | 1.58 (0.62)
Statistical Analysis 1: Comparison: Pulmonary Rehabilitation Group 6 Weeks FEV1,Liter(L)/Sec vs The Control Group 6 Weeks FEV1,Liter(L)/Sec; Test type: Superiority; p < 0.05, ANOVA

15. Secondary Outcome: Discharge 6weeks MMEF 25-75%(Liter(L)/Sec)
Description: as for outcome 6
Time Frame: assessed at discharge 6 weeks
Population: 2-WAY repeated measures ANOVA method was used for pulmonary function test.
Measure: Mean (Standard Deviation); unit: liter(L)/sec
Groups:
- Pulmonary Rehabilitation Group 6 Weeks MMEF(Liter(L)/Sec); The Control Group 6 Weeks MMEF(Liter(L)/Sec): Each subject received MMEF assessments at 6 weeks after discharge
Arm/Group | Pulmonary Rehabilitation Group 6 Weeks MMEF(Liter(L)/Sec) | The Control Group 6 Weeks MMEF(Liter(L)/Sec)
Number analyzed (Participants) | 18 | 18
liter(L)/sec | 2.12 (0.74) | 2.08 (1.46)
Statistical Analysis 1: Comparison: Pulmonary Rehabilitation Group 6 Weeks MMEF(Liter(L)/Sec) vs The Control Group 6 Weeks MMEF(Liter(L)/Sec); Test type: Superiority; p < 0.05, ANOVA

16. Secondary Outcome: Discharge 6weeks Peak Expiratory Flow Rate(PEFR in Liter( L)/Sec)
Description: as for outcome 7
Time Frame: assessed at discharge .6weeks
Population: 2-WAY repeated measures ANOVA method was used for pulmonary function test.
Measure: Mean (Standard Deviation); unit: liter(L)/sec
Groups:
- Pulmonary Rehabilitation Group: Each subject received PEFRassessments at 6 week after discharge
- The Control Group: Each subject received PEFR assessments at 6 weeks after discharge
Arm/Group | Pulmonary Rehabilitation Group | The Control Group
Number analyzed (Participants) | 18 | 18
liter(L)/sec | 5.13 (1.50) | 4.71 (2.13)
Statistical Analysis 1: Comparison: Pulmonary Rehabilitation Group vs The Control Group; null hypothesis; Test type: Superiority; p < 0.05, ANOVA

17. Secondary Outcome: Discharge 6 Weeks Inspiratory Muscle Strength(MIP,cmH2O)
Description: as for outcome 8
Time Frame: assessed at discharge6 weeks.
Population: Two-way repeated measures ANOVA for MIP. an intention-to-treat analysis was performed.group × time interactions were observed for the MIP
Measure: Mean (Standard Deviation); unit: cmH2O
Groups:
- Pulmonary Rehabilitation Group MIP(cmH2O); The Control Group MIP(cmH2O): Each subject received MIP assessments at discharge 6 weeks
Arm/Group | Pulmonary Rehabilitation Group MIP(cmH2O) | The Control Group MIP(cmH2O)
Number analyzed (Participants) | 18 | 18
cmH2O | 93.33 (34.47) | 64.67 (20.3)

18. Secondary Outcome: Discharge 6weeks Expiratory Muscle Strength (MEP, cmH2O)
Description: The Maximal Expiratory Pressure (MEP,cmH2O) are global measures of the maximal strength of the respiratory muscles.(MEP, cmH2O) .MEP is a supra-atmospheric pressure which can be developed in an effort of the abdominal and intercostal muscles.Expiratory muscle strength assesses extrathoracic muscle health.An absolute MEP value of < 80 cm H2O is always abnormal, and higher scores mean a better outcome.
Time Frame: assessed at discharge 6 weeks
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: cmH2O
Groups:
- Pulmonary Rehabilitation Group 6 Weeks MEP(cmH2O); The Control Group 6 Weeks MEP(cmH2O): Each subject received MEP assessments at discharge, and 2 weeks, 6 weeks, and 12 weeks after discharge
Arm/Group | Pulmonary Rehabilitation Group 6 Weeks MEP(cmH2O) | The Control Group 6 Weeks MEP(cmH2O)
Number analyzed (Participants) | 18 | 18
cmH2O | 93.89 (30.70) | 76.67 (23.51)
Statistical Analysis 1: Comparison: Pulmonary Rehabilitation Group 6 Weeks MEP(cmH2O) vs The Control Group 6 Weeks MEP(cmH2O); Test type: Superiority; p < 0.05, ANOVA

19. Secondary Outcome: Discharge 6 Weeks Modified Borg Score
Description: as for outcome 10
Time Frame: assessed at discharge 6week
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- Pulmonary Rehabilitation Group 6 weeksModified Borg Score; The Control Group 6 Weeks Modified Borg Score: Each subject received Modified Borg score assessments at discharge, and 2 weeks, 6 weeks, and 12 weeks after discharge
Arm/Group | Pulmonary Rehabilitation Group 6 weeksModified Borg Score | The Control Group 6 Weeks Modified Borg Score
Number analyzed (Participants) | 18 | 18
scores on a scale | 0.75 (0.79) | 1.11 (1.74)
Statistical Analysis 1: Comparison: Pulmonary Rehabilitation Group 6 weeksModified Borg Score vs The Control Group 6 Weeks Modified Borg Score; Test type: Superiority; p < 0.05, ANOVA

20. Secondary Outcome: Discharge 6weeks Lung Expansion Capacity
Description: Lung expansion capacity as assessed by incentive spirometry with the flow-oriented device( Triflow II,volume × seconds) (ml)).Incentive spirometry that feedback respiratory training can improve respiratory function, endurance for exercise capacity,Wide flow rate range from 600 - 1200(volume × seconds) (mL)c.higher scores mean a better outcome.
Time Frame: assessed at discharge 6 weeks
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: (ml)
Groups:
- Pulmonary Rehabilitation: study group follow incentive spirometry with the flow-oriented device( Triflow II,(cc/sec) on discharge 6 weeks
- Control Group: control group follow incentive spirometry with the flow-oriented device( Triflow II,(cc/sec) on discharge 6 weeks
Arm/Group | Pulmonary Rehabilitation | Control Group
Number analyzed (Participants) | 18 | 18
(ml) | 1683.33 (667.96) | 1116.63 (382.33)
Statistical Analysis 1: Comparison: Pulmonary Rehabilitation vs Control Group; Test type: Superiority; p < 0.05, ANOVA

21. Secondary Outcome: Postoperative 6weeks Pulmonary Complications
Description: Pulmonary complication as assessed by Chest X-ray.pneumonia.lung collapse.atelectasis.emphysema and pleural effusion were collected.In our research,some patients have two pulmonary complications at the same time, such as emphysem and infiltration, so the total number is not necessarily equal to 18.
Time Frame: at 6weeks after discharge
Population: Pearson chi-square test was used for Pulmonary complication on discharge 6 weeks .Data is presented as n(%).
Measure: Count of Participants; unit: Participants
Groups:
- Pulmonary Rehabilitation: study group follow CXR on discharge 6 weeks
- Control Group: control group follow CXR on discharge 6 weeks
Arm/Group | Pulmonary Rehabilitation | Control Group
Number analyzed (Participants) | 18 | 18
Participants
  pneumonia | 0 | 1
  atelectasis | 0 | 2
  pleural effusion | 3 | 4
  emphysema | 5 | 11
  pulmonary infilation | 1 | 1
Statistical Analysis 1: Comparison: Pulmonary Rehabilitation vs Control Group; null hypothesis; Test type: Superiority; p < 0.05, Chi-squared

22. Secondary Outcome: Discharge 12 Weeks Forced Vital Capacity (FVC in Liter(L)/Sec )
Description: as for outcome 13
Time Frame: assessments at discharge 12 weeks
Population: .2-WAY repeated measures ANOVA method was used for pulmonary function test.
Measure: Mean (Standard Deviation); unit: liter( L)/sec
Groups:
- Pulmonary Rehabilitation Group; The Control Group: Each subject received FVC(L/sec) assessments at 12 weeks after discharge
Arm/Group | Pulmonary Rehabilitation Group | The Control Group
Number analyzed (Participants) | 18 | 18
liter( L)/sec | 2.32 (0.72) | 2.16 (0.96)
Statistical Analysis 1: Comparison: Pulmonary Rehabilitation Group vs The Control Group; null hypothesis; Test type: Superiority; p < 0.05, ANOVA

23. Secondary Outcome: Discharge 12 Weeks Forced Expiratory Volume in 1 Second(FEV1,Liter(L)/Sec)
Description: The Forced Expiratory Volume in 1 Second parameter(FEV1,liter(L)/sec) measures the volume of air that was exhaled into the mouthpiece in the first second after a full inhalation. The Measured column represents the total volume exhaled during the first second, in liters. Normal values in healthy males aged 20-60 range from 4.5 to 3.5 liters, and normal values for females aged 20-60 range from 3.25 to 2.5 liters. The Predicted column compares the actual volume breathed out during the first second of your test to an average of the normal volume breathed out in 1 second for a person of the same gender, height, and age. This value is expressed as a percentage, with normal test values being between 80% and 120% of the average (predicted) values.and whether higher scores mean a better outcome.
Time Frame: assessed at discharge12weeks
Population: 2-WAY repeated measures ANOVA method was used for pulmonary function test.
Measure: Mean (Standard Deviation); unit: liter(L)/sec
Groups:
- Pulmonary Rehabilitation Group 12 Weeks FEV1,Liter(L)/Sec; The Control Group 12 Weeks FEV1,Liter(L)/Sec: Each subject received FEV1 assessments at discharge12 weeks after discharge
Arm/Group | Pulmonary Rehabilitation Group 12 Weeks FEV1,Liter(L)/Sec | The Control Group 12 Weeks FEV1,Liter(L)/Sec
Number analyzed (Participants) | 18 | 18
liter(L)/sec | 1.85 (0.45) | 1.74 (0.72)
Statistical Analysis 1: Comparison: Pulmonary Rehabilitation Group 12 Weeks FEV1,Liter(L)/Sec vs The Control Group 12 Weeks FEV1,Liter(L)/Sec; null hypothesis; Test type: Superiority; p < 0.05, ANOVA

24. Secondary Outcome: Discharge 12 Weeks MMEF 25-75%(Liter(L)/Sec)
Description: as for outcome 6
Time Frame: assessed at discharge12weeks "
Population: 2-WAY repeated measures ANOVA method was used for pulmonary function test.
Measure: Mean (Standard Deviation); unit: liter(L)/sec
Groups:
- Pulmonary Rehabilitation Group 12weeks MMEF(Liter(L)/Sec); The Control Group 12 Weeks MMEF(Liter(L)/Sec): Each subject received MMEF assessments at 12 weeks after discharge
Arm/Group | Pulmonary Rehabilitation Group 12weeks MMEF(Liter(L)/Sec) | The Control Group 12 Weeks MMEF(Liter(L)/Sec)
Number analyzed (Participants) | 18 | 18
liter(L)/sec | 2.44 (1.50) | 1.85 (0.76)
Statistical Analysis 1: Comparison: Pulmonary Rehabilitation Group 12weeks MMEF(Liter(L)/Sec) vs The Control Group 12 Weeks MMEF(Liter(L)/Sec); Test type: Superiority; p < 0.05, ANOVA

25. Secondary Outcome: Discharge 12 Weeks Peak Expiratory Flow Rate (PEFR in Liter(L)/Sec)
Description: as for outcome 7
Time Frame: assessed at discharge 12 weeks
Population: 2-WAY repeated measures ANOVA method was used for pulmonary function test.
Measure: Mean (Standard Deviation); unit: liter(L)/sec
Groups:
- Pulmonary Rehabilitation Group; The Control Group: Each subject received PEFR assessments at 12 weeks after discharge
Arm/Group | Pulmonary Rehabilitation Group | The Control Group
Number analyzed (Participants) | 18 | 18
liter(L)/sec | 4.94 (1.46) | 4.78 (2.25)
Statistical Analysis 1: Comparison: Pulmonary Rehabilitation Group vs The Control Group; null hypothesis; Test type: Superiority; p < 0.05, ANOVA

26. Secondary Outcome: Discharge 12 Weeks Inspiratory Muscle Strength (MIP,cmH2O)
Description: as for outcome 8
Time Frame: assessed at discharge12 weeks.
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: cmH2O
Groups:
- Pulmonary Rehabilitation Group; The Control Group(MIP,cmH2O): Each subject received MIP assessments at discharge 12 weeks
Arm/Group | Pulmonary Rehabilitation Group | The Control Group(MIP,cmH2O)
Number analyzed (Participants) | 18 | 18
cmH2O | 91.11 (30.46) | 64.67 (20.30)

27. Secondary Outcome: Discharge 12weeks Expiratory Muscle Strength(MEP,cmH2O)
Description: as for outcome 18
Time Frame: assessed at discharge 12weeks
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: cmH2O
Groups:
- Pulmonary Rehabilitation Group 12 Weeks MEP(cmH2O); The Control Group 12 Weeks MEP(cmH2O): Each subject received MEP assessments at discharge, and 2 weeks, 6 weeks, and 12 weeks after discharge
Arm/Group | Pulmonary Rehabilitation Group 12 Weeks MEP(cmH2O) | The Control Group 12 Weeks MEP(cmH2O)
Number analyzed (Participants) | 18 | 18
cmH2O | 92.56 (34.37) | 74.48 (18.64)
Statistical Analysis 1: Comparison: Pulmonary Rehabilitation Group 12 Weeks MEP(cmH2O) vs The Control Group 12 Weeks MEP(cmH2O); Test type: Superiority; p < 0.05, ANOVA

28. Secondary Outcome: Discharge 12 Weeks Modified Borg Score
Description: as for outcome 10
Time Frame: assessed at discharge12weeks
Population: Two-way repeated measures ANOVA for Modified Borg score. an intention-to-treat analysis was performed.group × time interactions were observed for the Modified Borg score
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- Pulmonary Rehabilitation Group 12weeksModified Borg Score; The Control Group 12 Weeks Modified Borg Score: Each subject received Modified Borg score assessments at discharge, and 2 weeks, 6 weeks, and 12 weeks after discharge
Arm/Group | Pulmonary Rehabilitation Group 12weeksModified Borg Score | The Control Group 12 Weeks Modified Borg Score
Number analyzed (Participants) | 18 | 18
scores on a scale | 0.70 (0.83) | 1.05 (0.92)
Statistical Analysis 1: Comparison: Pulmonary Rehabilitation Group 12weeksModified Borg Score vs The Control Group 12 Weeks Modified Borg Score; Test type: Superiority; p < 0.05, ANOVA

29. Secondary Outcome: Discharge 12 Weeks Lung Expansion Capacity
Description: as for outcome 20
Time Frame: assessed at discharge 12weeks
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: (ml)
Groups:
- Pulmonary Rehabilitation: study group follow incentive spirometry with the flow-oriented device( Triflow II,(cc/sec) on discharge12 weeks
- Control Group: control group follow incentive spirometry with the flow-oriented device( Triflow II,(cc/sec) on discharge12 weeks
Arm/Group | Pulmonary Rehabilitation | Control Group
Number analyzed (Participants) | 18 | 18
(ml) | 1406.67 (798.20) | 1150.33 (345.13)
Statistical Analysis 1: Comparison: Pulmonary Rehabilitation vs Control Group; Test type: Superiority; p < 0.05, ANOVA

30. Secondary Outcome: Postoperative 12 Weeks Pulmonary Complications
Description: as for outcome 12
Time Frame: at 12 weeks after discharge
Population: Pearson chi-square test was used for Pulmonary complication on discharge 12 weeks .Data is presented as n(%).
Measure: Count of Participants; unit: Participants
Groups:
- Pulmonary Rehabilitation: study group follow CXR on discharge12 weeks
- Control Group: control group follow CXR on discharge 12 weeks
Arm/Group | Pulmonary Rehabilitation | Control Group
Number analyzed (Participants) | 18 | 18
Participants
  pneumonia | 0 | 1
  atelectasis | 1 | 2
  pleural effusion | 0 | 1
  emphysema | 1 | 0
  pulmonary infilation | 0 | 1

ADVERSE EVENTS:
Time Frame: we collect 12 weeks of adverse event data
Description: Before discharge,If air leakage occurs before discharge, we definition it as an adverse event, because it may extend the patient's hospital stay.After discharge, home-based rehabilitation program design as a low-to-medium intensity and non-invasive .Researchers contacted patients at home every week through phone calls to monitor the occurrence of any uncomfortable reaction and post-op 2weeks,6weeks and 12weeks regular check CXR .PFT. 6min walking test and respiratory muscle power .
Groups:
- Pulmonary Rehabilitation Group: 0-2 weeks, the aerobic exercise intensity was targeted to reach 10-11 points of RPE scale. Patients raised their upper limbs while simultaneously performing lower-limb stepping at place for 20 min; in addition, they walked at a comfortable speed for 15 min twice per day.Triflo-II was performed 8-10 times per hour. inspiratory muscle training (30 breaths each time, twice per day) with the initial pressure set at 25%-30% of the maximum inspiratory pressure.
  3-6 weeks, the aerobic exercise intensity was targeted to reach 12-15 points on the RPE scale. Patients performed upper-limb resistance exercise (raising of a 250-cc water bottle) and lower-limb stepping for 20 min per day as well as walking exercise (slow walking for 5 min and fast walking for 2 min, followed by 5-min slow walking, for a total of 30 min).Triflo-II was performed 8-10 times per hour, and inspiratory muscle training, with the pressure intensity adjusted to more than 5% of that in the first stage.
- The Control Group: The control group accept the pulmonary rehabilitation , breathing exercise, extremities exercise, breathing muscle training, incentive spirometry (Triflo-II) training, intermittent positive pressure ventilation, chest physical therapy and pain control) only in operation stage on before op-day 3 day and after op-day and without home based pulmonary rehabilitation.
Arm/Group | Pulmonary Rehabilitation Group | The Control Group
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 6/18 | 6/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pulmonary Rehabilitation Group (N=18) | The Control Group (N=18)
Prolonged air leak (PAL) (Surgical and medical procedures) | 6 (18) | 6 (18) — Prolonged air leak (PAL) is one of the most common postoperative complications after pulmonary resection Pleural adhesion was associated with increased risk of PAL ,and will prolong hospital stay after surgery.

LIMITATIONS AND CAVEATS:
First,sample size is low,this may affect the result of the study;secondly, pulmonary function should collect DLCO and MVV;third,although the patients were checked via telephone every week,there is no surefire way to enforce intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-31): https://cdn.clinicaltrials.gov/large-docs/92/NCT02757092/Prot_SAP_000.pdf